CLINICAL TRIAL: NCT06826378
Title: Observational Study Between Patients Undergoing Total Intracorporeal Anastomosis Or Extracorporeal Anastomosis After Segmental Resection For Deep Endometriosis
Brief Title: Patients Undergoing Total Intracorporeal or Extracorporeal Anastomosis After Segmental Resection for Deep Endometriosis
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ARISTOTLE23
Record Dates: First submitted 2024-12-03; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-10

CONDITIONS: Deep Endometriosis
Keywords: Endometriosis; Gynaecology; Surgery; Anastomosis; Segmental resection
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Impact on the quality of life (in terms of functional recovery and gastrointestinal symptoms) of segmental resection surgery in patients with intestinal endometriosis undergoing either a totally intracorporeal or extracorporeal procedure

DETAILED DESCRIPTION:
Surgery is the treatment of choice for deep endometriosis with bowel involvement and endometriosis nodules will be treated by segmental resection and subsequent anastomosis packing. Anastomosis packing with a totally intracorporeal approach may be a successful solution to reduce some of the complications after discoid or segmental resection with conventional laparotomic approach for extracorporeal anastomosis.

Setting up the colorectal anastomosis with a totally intracorporeal approach represents a surgical method that has been recently introduced but is already approved in terms of safety and reproducibility. However, experience with this technique is currently limited and there is no established consensus regarding patient suitability or data on longer-term outcomes. New studies are therefore needed to further validate the technique and to fully assess its long-term benefits resulting in increased quality of life for operated patients or to identify any associated complications.

The aim of the study is therefore to describe the impact on the quality of life (in terms of functional recovery and gastrointestinal symptoms) of segmental resection surgery in patients with intestinal endometriosis who underwent either a totally intracorporeal or extracorporeal procedure. In addition, the aim is to detect any differences in the duration of the operating time, compare the duration of the postoperative hospital stay and determine the success rate of the totally intracorporeal procedure

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 54 years of age
* Diagnosis, by instrumental examination such as transvaginal ultrasound, of deep endometriosis with suspected intestinal involvement
* Intraoperative indication for segmental resection for intestinal endometriosis
* Obtaining informed consent for study participation and data processing

Exclusion Criteria:

* Patients with a known concomitant inflammatory bowel syndrome (inflammatory bowel syndrome)
* Patients undergoing emergency/emergency surgery

Ages: 18 Years to 54 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with deep endometriosis with suspected bowel involvement and intraoperative indication for segmental resection
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Impact on the quality of life (in terms of functional recovery and gastrointestinal symptoms) of segmental resection surgery in patients with intestinal endometriosis undergoing either a totally intracorporeal or extracorporeal procedure | During the preoperative evaluation and at 3 months after surgery as part of the postoperative follow-up visit
  Evaluation by scoring the validated Low Anterior Resection Syndrome score questionnaire

SECONDARY OUTCOMES:
Detect any differences in the duration of the total operating time in the two different treatments | During surgery
  Total operating time measured in minutes
Duration of hospitalisation in the two different types of surgery | From date of surgery until the discharge (0-30 days)
  Measurement of hospitalisation time after surgery
Success rate of the totally intracorporeal procedure in patients with deep endometriosis with bowel involvement undergoing segmental resection surgery | At 3 months after surgery
  Number of successfully completed operations out of the total number of operations performed with a fully intracorporeal approach. The success of the intervention is established intraoperatively by performing hydropneumatic tests of the integrity of the anastomosis and during the operative course by assessing the possible occurrence of complications
Incidence of intra-operative complications (rectorrhagia, anastomotic dehiscence, intussusception, stenosis of the anastomosis, intraperitoneal haemorrhage, conversion to laparotomic surgery) and evaluate any differences in these between the two groups | At 3 months after surgery
  Number of operations in which one (or more) of the intra-operative complications occurred out of the total number of operations performed with a totally intracorporeal approach
Incidence of post-operative complications in the two different surgical treatments | Within 3 months of surgery
  Number of operations in which one (or more) of the post-operative complications described above occurred out of the total number of operations performed

CONTACTS AND LOCATIONS:
Overall Officials: Diego Raimondo, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy